CLINICAL TRIAL: NCT05745636
Title: Influence of TrueBroc® Broccoli Seed Extract Supplementation on Skin Health
Brief Title: Broccoli Seed Extract and Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: North Carolina State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HS-22-42
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-06

CONDITIONS: Skin Inflammation
Keywords: broccoli; Glucoraphanin; inflammation; skin; sulforaphane (
MeSH Terms: conditions — Dermatitis; Inflammation | interventions — Amines; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, crossover design with 4-week supplementation periods and a 2-week washout period.
Who Masked: Participant, Investigator
Masking Description: Experimental and placebo capsules (2 consumed per day for 4 weeks) will look identical. Both the investigators and the subjects will be blinded, with the code held by the sponsor until the study and data analysis have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broccoli, mustard, vitamin C (Experimental): 770 mg Broccoli Seed Extract (BSE) with 290 mg mustard seed powder (MSP) and 200 mg vitamin C
  Interventions: Dietary Supplement: Broccoli, mustard, vitamin C
- Placebo (Placebo Comparator): inactive excipients including microcrystalline cellulose, rice hull, maltodextrin, ascorbyl palmitate and silicon dioxide
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Broccoli, mustard, vitamin C — 2 capsules per day for 4 weeks
  Arms: Broccoli, mustard, vitamin C
Dietary Supplement: Placebo — 2 capsules per day for 4 weeks.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to examine the influence of 4-weeks ingestion of TrueBroc®, (broccoli seed extract, BSE) with mustard seed powder (MSP) on improving skin health by evaluating skin physiological and biochemical parameters. This study will test the effect of BSE and MSP compared to placebo on skin health after 4 weeks supplementation. The study will employ a randomized, crossover design with subjects acting as their own controls.

DETAILED DESCRIPTION:
The primary objective of this study is to examine the influence of 4-weeks ingestion of TrueBroc® with mustard seed powder on improving skin health by evaluating skin physiological and biochemical parameters. TrueBroc® Glucoraphanin-Rich Broccoli Seed Extract (TrueBroc®) is a hot water extract of Brassica oleracea var. Italica Plenck (Brassicaceae) seeds. TrueBroc® contains high levels of glucoraphanin, a glucosinolate prominently found in the cruciferous vegetables. This study will use supplements containing 770 mg Broccoli Seed Extract (BSE) with 290 mg mustard seed powder (MSP) and 200 mg vitamin C. Limited data indicate that this mixture enhances glucoraphanin bioavailability. The consumption of the phytochemical glucoraphanin confers a number of benefits including skin health.

Hypothesis: That 4-weeks ingestion of TrueBroc® with MSP compared to placebo will improve skin health.

Study Procedures This study will incorporate a randomized, double-blinded, placebo-controlled, crossover design with 4-week supplementation and a 2-week washout period. Skin measurements and tape stripping samples will be collected pre- and post-4-week supplementation periods. Skin tape stripping samples will be analyzed for oxinflammatory-related outcomes. Blood and 24-hour urine samples will also be collected pre- and post-4-week supplementation periods. These samples will be aliquoted and stored in a freezer for potential analysis of targeted outcomes pending additional funding.

Visit #1: Screening and Consent. Subjects will come to the Human Performance Lab at assigned times. The COVID-19 screening participant form will be filled in by the participant to verify the absence of symptoms or exposure.This visit will begin with a review of the consent form, and the inclusion and exclusion criteria. Height, body weight, body composition (seca BIA), and blood pressure will be measured. Subjects will be given 24-hour collection kits with instructions to collect all urine in the provided jug during the day before visit #2.

Visit #2: Return urine bottles. Provide blood sample. Skin health measurements. Start 4-weeks supplementation.

Subjects will come to the Human Performance Lab at assigned times in an overnight fasted state (no intake of food or beverages except for water during at least the previous 9 hours). Subjects will drop off the urine bottles and provide an overnight fasted blood sample. Skin health measurements will involve having probes and tapes applied to the surface of the skin to assess various parameters of skin health. Photos of skin areas will be taken. These skin health measurements will take about 15 to 30 minutes. A 4-week supply of capsules will be provided in supplement trays or bottles, and an additional 24-hour urine collection kit will be given to each subject. Subjects will be contacted weekly by the Research Manager to ensure adherence to the supplementation regimen (2 capsules per day, 4 weeks). Visit #3: Repeat visit #2 test procedures. Subjects will come to the Human Performance Lab at assigned times in an overnight fasted state after 4 weeks of supplementation. Subjects will drop off the urine bottles and provide a blood sample. Body composition and blood pressure measurements will be repeated. Skin health measurements will be repeated. An additional 24-hour urine collection kit will be given to each subject. Subjects will be instructed to return to the lab after the 2-week washout period.

Visits #4 and #5: Repeated procedures from visits #2 and #3. Subjects will crossover to the opposite trial supplement and repeat all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects will be included, ages 25 to 57 years.
* Non-smoker and free of any medical conditions that might affect study measurements.
* Body mass index (BMI) of 20 - 29.9 kg/m2 (not obese).
* Willingness to adhere to dietary restrictions: refrain from consuming cruciferous vegetables (or related condiments and supplements) such as broccoli, cauliflower, cabbage, kale, bok choy, arugula, Brussels sprouts, collards, watercress, radishes, prepared mustard condiment, mustard greens, horseradish, wasabi, and mayonnaise for 3 days before and for the duration of the study.
* Willing to collect all urine for 24 hours and provide four blood samples on four separate occasions.

Exclusion Criteria:

* Diarrhea or oral antibiotic intake within the last 4 weeks.
* Use of proton pump inhibitors (PPIs), antacids or other medications that influence stomach acidity.
* History of malabsorption or GI tract disorders or GI surgeries (i.e. lapband, gastric bypass, etc.).
* History of allergic reactions or intolerance to any of the ingredients contained in the test supplements (e.g. broccoli, broccoli seeds, mustard seeds, vitamin C).
* Currently pregnant, planning to become pregnant, or breastfeeding.
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 25 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Skin IL-1beta (pg/ml) | Change from pre-study to post-4 weeks supplementation
  Skin inflammation cytokine

SECONDARY OUTCOMES:
Skin elasticity (arbitrary units) | Change from pre-study to post-4 weeks supplementation
  DermaLab® Combo elasticity probe measurement
Skin pH (arbitrary units) | Change from pre-study to post-4 weeks supplementation
  DermaLab® Combo pH probe measurement
Skin hydration (arbitrary units) | Change from pre-study to post-4 weeks supplementation
  DermaLab® Combo hydration probe measurement
Skin pigmentation (melatonin content, no units) | Change from pre-study to post-4 weeks supplementation
  DermaLab Combo color probe
Transepidermal water loss (TEWL) (g/m2/h) | Change from pre-study to post-4 weeks supplementation
  DermaLab® Combo TEWL probe measurement
Skin sebum (arbitrary units) | Change from pre-study to post-4 weeks supplementation
  DermaLab® Combo sebum probe measurement

CONTACTS AND LOCATIONS:
Overall Officials: Camila A Olson, PhD, Study Director — Appalachian State University
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States